CLINICAL TRIAL: NCT00896415
Title: Inter-scanner Comparison of Muscle Attenuation Measures
Brief Title: Interscanner Variation in Musculoskeletal Computed Tomography (CT) Measures
Acronym: Interscanner
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Thomas Lang, PhD Professor in Residence, Department of Radiology, University of California San Francisco
Other Study IDs: Inter-scanner study; TLANG_Interscanner
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2009-05

CONDITIONS: Accidental Falls; Loss of Muscle Strength
Keywords: on two models of CT scanner acquire CT images of the abdomen pelvis and midthigh in 20 Postmenopausal female volunteers

STUDY DESIGN:
Observational Model: Ecologic or Community

SUMMARY:
Maintaining strong muscles is important for the independence and quality of life in our older population. Strong muscles provide mobility and reduce the chance of falls that lead to injury. Many researchers are carrying out studies to examine different types of exercise and drug treatments to prevent loss of muscle strength in older people. Often, these research studies use x-ray computed tomography (CT) scans to measure the size and the amount of fat in different muscles. These factors are known to reflect muscle health. Large studies can involve many research subjects recruited at many different clinics with different CT scanners. To ensure that these studies provide reliable results, the investigators must have procedures to make sure that different CT scanners measure the same results for the same amount of fat or muscle. The goal of our study is to develop these procedures. In this project, the investigators will study women because they have the highest risk of bone fractures resulting from falls. Thus, the subjects are being asked to volunteer for a study where the subjects will be scanned on different scanners.

ELIGIBILITY:
Inclusion Criteria:

* age 60-70 years old
* healthy

Exclusion Criteria:

* no history of spine surgery
* no history of hip implantation or replacement
* no scoliosis or other spine deformity
* not using walking canes or wheelchair

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this project we will study women 60-70 years old because they have the highest risk of bone fractures resulting from falls.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-05; Study Completion 2009-11 (Actual)